CLINICAL TRIAL: NCT06587438
Title: Effects of COntinuous Glucose MoNitoring Versus Usual Care on GlycEmic Control in Non-insulin-tReated Adults with Type 2 Diabetes：a Multi-center Randomized Controlled Trial
Brief Title: Effect of CGM on Glucose Control in Non-insulin-treated Patients with Type 2 Diabetes Mellitus
Acronym: CONVERT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinocare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SN-CGM-PO-001
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real-time Continuous glucose monitor (Experimental): In the first two weeks of every four-week period, rt-CGM is used to monitor blood glucose levels, while in the latter two weeks, SBMG is employed for usual care
  Interventions: Device: Sinocare iCan I3 CGM
- Self-monitoring of blood glucose (Active Comparator): Using SMBG for usual care only.
  Interventions: Device: Sinocare jinzhi+Blood glucose meter

INTERVENTIONS:
Device: Sinocare iCan I3 CGM — Real-time Continuous glucose monitoring
  Arms: Real-time Continuous glucose monitor
Device: Sinocare jinzhi+Blood glucose meter — Self-monitoring of blood glucose
  Arms: Self-monitoring of blood glucose

SUMMARY:
The clinical value of CGM for diabetic patients undergoing insulin therapy has been widely recognized, but the evidence-based support for its use in non-insulin-treated type 2 diabetic patients remains insufficient. The primary objective of this study is to evaluate the effect of real-time continuous glucose monitoring (CGM) compared with self-monitoring of blood glucose on glycemic control in adults with non-insulin treated type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* (1)Subjects aged ≥18 years at screening (based on the day of signing the informed consent form) and of any gender
* (2)Patients diagnosed with type 2 diabetes
* (3)Prior to the screening, glycemic control was suboptimal with diet, exercise control, and oral medication or glucagon-like peptide-1RA (GLP-1RA) therapy maintained for more than 3 months, 7.5%≤HbA1c≤10%
* (4)Subjects voluntarily sign an informed consent form

Exclusion Criteria:

* (1)Patients treated with insulin within 3 months prior to screening
* (2)Currently or have used a CGM device within 3 months prior to enrollment
* (3)Serious skin disease at the sensor placement site, allergy to tape or adhesives
* (4)Pregnant females, those with a positive pregnancy test result at screening, or those who plan to become pregnant during the study
* (5)Those who are participating or will participate in other clinical trials
* (6)Those who, in the opinion of the investigator, should not participate in this clinical trial, such as: ①those who have a history of eye trauma or other diagnosed eye diseases resulting in visual impairment, etc.; ②those who are unwilling or unable to fully understand or cooperate due to speech disorders; ③those who suffer from mental disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 24 weeks
  Between group differences (CGM and SMBG) for the change in HbA1c (from Central Lab) from baseline to week 24.

IPD SHARING:
Plan to Share IPD: No